CLINICAL TRIAL: NCT03360240
Title: Levels of Blood Pressure in Adolescents With Preclampsia and Eclampsia: Study of Cases and Controls.
Brief Title: Blood Pressure in Adolescents With PReclampsia and Eclampsia.
Acronym: ADPRE
Status: Completed | Type: Observational
Sponsor: Complejo Hospitalario Dr. Arnulfo Arias Madrid (Other)
Responsible Party: Principal Investigator, Paulino Vigil-De Gracia, Gynecology and Obstetric, Complejo Hospitalario Dr. Arnulfo Arias Madrid
Other Study IDs: Latin Adolescents
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Adolescent Pregnancy; Preeclampsia and Eclampsia
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 11 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases: patients with pregnancy that starts before the age of 19 that develops preeclampsia (mild), severe preeclampsia, gestational hypertension and eclampsia, that is 24 and more weeks pregnant with prenatal control started before 20 weeks of pregnancy.
- controls: Are patients with pregnancy that starts before the age of 19 that without develops (preeclampsia mild), severe preeclampsia, gestational hypertension or eclampsia) that is 24 and more weeks pregnant with prenatal control started before 20 weeks of pregnancy.

SUMMARY:
Levels of blood pressure in adolescents with preeclampsia and eclampsia:

Multicenter case-control study (Latin America). Maternities in Latin America: Two hospitals in Panama, one hospital in Mexico, one hospital in El Salvador, one hospital in Guatemala, two hospitals in Honduras, one hospital in Colombia, two hospitals in Peru and two hospitals in Bolivia.

The objective is to evaluate the basal levels of blood pressure during pregnancy and determine if there is any increase that is associated with the development of preeclampsia and eclampsia without reaching the known values of 140/90 mm Hg.

The sample is 1050: (350 Cases and 700 Controls).

DETAILED DESCRIPTION:
Levels of blood pressure in adolescents with preeclampsia and eclampsia: cases and controls study.

It is unknown whether the blood pressure levels used for the diagnosis of preeclampsia have the same impact in adolescents as in older women, however for the diagnosis of preeclampsia and severe hypertension the same criteria of hypertension are used regardless of age maternal.

It is necessary to do research to determine the values of blood pressure with which adolescents convulse and also to validate if slight increases in baseline blood pressure in adolescents are associated with prediction of preeclampsia and eclampsia.

Unfortunately, 85% of teenage pregnancies occur in non-industrialized countries such as those in Latin America, and it is estimated that 25% of maternal deaths occur in adolescents

Cases: patients with pregnancy that starts before the age of 19 that develops preeclampsia (mild), severe preeclampsia, gestational hypertension and eclampsia, that is 24 and more weeks pregnant with prenatal control started before 20 weeks of pregnancy. Controls are patients with the same criteria but WITHOUT hypertension during this pregnancy.

The statistical analyzes are based on comparing blood pressure levels between the two groups, in addition blood pressure levels like 30/15 on the systolic and diastolic basal levels will be created and compared between the two groups, especially when it is not possible to have 140 / 90 mm Hg.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion cases: Patients with pregnancy that starts before the age of 19 that develops preeclampsia (mild), severe preeclampsia, gestational hypertension and eclampsia, that has 24 and more weeks of pregnancy with prenatal control started before 20 weeks of age. pregnancy. That you get the data of the termination of your pregnancy.

Exclusion Criteria:

* Patients with pregnancy that starts before 19 years of age that does NOT develop preeclampsia (mild), severe preeclampsia, gestational hypertension and eclampsia, that has 24 and more weeks of pregnancy with prenatal control started before 20 weeks of pregnancy. That you get the data of the termination of your pregnancy.

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant patients who are 19 years of age or younger and more than 23 weeks pregnant, where the cases are those that develop preeclampsia (mild), severe preclampsia, gestational hypertension and eclampsia; and the controls patients of the same age and with more than 23 weeks of pregnancy without hypertension.
Sampling Method: Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Levels of blood pressure | after 24 weeks of gestactión to delivery.
  Level of blood pressure during pregnancy or delivery

SECONDARY OUTCOMES:
severe hypertension | after 24 weeks of gestactión to delivery.
  hypertension more thet 160 mmHg on systolic or 110 mmHg on diastolyc.
parity | birth before actual pregancy
  number of previous birth

CONTACTS AND LOCATIONS:
Overall Officials: Paulino Vigil, Principal Investigator — Complejo CSS
Locations (8):
- Hospital del seguridad social La Paz, La Paz, Bolivia
- Hospital de Pereira, Pereira, Colombia
- Hospital de IGSS, Guatemala, Guatemala City, Guatemala
- Hospial de Honduras, Tegucigalpa, Honduras
- Panama (2):
  - Complejo Hospitalario CSS, Panama City
  - Santo Tomás, Panama City
- Peru (2):
  - Hospital Regional de Cajamarca, Cajamarca
  - Hospital Nacional Docente Madre Niño, San Bartolomé,, Lima

IPD SHARING:
Plan to Share IPD: No